CLINICAL TRIAL: NCT02312375
Title: Effects of Fimasartan on Insulin Secretion, and Interaction With DPP4 Inhibitors in Patients With Type 2 Diabetes
Brief Title: Effects of Fimasartan on Insulin Secretion in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hye Seung Jung, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Fimasartan study
Record Dates: First submitted 2014-12-03; First posted 2014-12-09 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fimasartan (Experimental): Expreimental drug is fimasartan.
  Interventions: Drug: Fimasartan
- Amlodipine (Active Comparator): Active comparator is amlodipine.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Fimasartan — 16 weeks of fimasartan vs. amlodipine followed by 2 weeks of wash-out period, then crossover
  Arms: Fimasartan
Drug: Amlodipine — 16 weeks of fimasartan vs. amlodipine followed by 2 weeks of wash-out period, then crossover
  Arms: Amlodipine

SUMMARY:
This study was designed to evaluate the effect of ARB in improving insulin secretion in patients with type 2 diabetes. The investigators also aimed to evaluate if there are potential synergisms between ARB and DPP4 inhibitors in improving insulin secretion and urinary albumin secretion in diabetic patients.

DETAILED DESCRIPTION:
Angiotensin II has been reported to insulin secretion in beta cells. Angiotensin II indirectly improves insulin secretion in beta cells via vasoconstriction and reduced islet blood flow. Chronic exposure to high glucose or high fat increases expression of AT1R (angiotensin type 1 receptor), leading to reactive oxidative stresses, inflammation, and apoptosis in beta cells, finally decreased insulin formation and secretion. Some studies showed the beneficial effect of blocking AT1R on insulin secretion and beta cell proliferation in animal models using angiotensin receptor blocker (ARB). Furthermore, 26 weeks of valsartan treatment improved insulin secretion in humans with impaired glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20~80 years
* Type 2 diabetic patients diagnosed more than 6 months ago
* HbA1c ≤8.5% at screening
* No change of OAD within the 3 months before screening
* SBP <140 mmHg and DBP <90 mmHg with anti-hypertensive drug at screening
* SBP ≥140 mmHg or DBP ≥80 mmHg without anti-hypertensive drug at screening

Exclusion Criteria:

* Type 1 diabetic patients or active insulin treatment at screening
* Treatment with ARB or ACEi within 1 month prior to screening
* Uncontrolled hypertension with SBP >170 mmHg or DBP >100 mmHg
* Pregnancy or lactation
* Elevated liver enzyme (AST or ALT > 3 times the UNL) or elevated serum Cr (≥1.5 mg/dL in men and 1.4 mg/dL in women)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Insulinogenic index | 16 week

SECONDARY OUTCOMES:
HOMA β-cell function | 16 week
Insulin resistance | 16 week
Urinary albumin creatinine ratio, urinary protein creatinine ratio | 16 week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea